CLINICAL TRIAL: NCT00526578
Title: Pancreatic Cancer Genetic Epidemiology (PACGENE) Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ID02-139; 1R01CA097075-01 (NIH)
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Pancreatic Cancer Genetic Epidemiology; PACGENE; Healthy Control; Familial Pancreatic Cancer; FPC; Questionnaire
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic carcinoma, familial | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Pancreatic cancer patients or family member.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire taking about 30-40 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this research study is to investigate the role of genes that may point to a higher risk of developing pancreatic cancer.

DETAILED DESCRIPTION:
Participants in this study will be part of a pancreatic cancer genetic epidemiology consortium (herein referred to as "PACGENE"), which includes researchers at these institutions: Mayo Clinic; Johns Hopkins University; Creighton University; University of Toronto Mount Sinai Hospital; Dana Farber; and Karmanos Cancer Institute. Participants have either been diagnosed with pancreatic cancer or are family members of pancreatic cancer patients.

Participants will be asked questions by a trained interviewer using an approved questionnaire. The topics will include demographic data (age, race, etc.), exposures, medical history data, family history of cancer and other conditions, and other lifestyle factors. It should take about 30-40 minutes to complete the questionnaire.

Participants in this study will also have about one and a half tablespoons of blood drawn. Blood that is collected will only be used by researchers involved in this study. If obtaining a blood sample is not possible, the study staff will ask for a saliva sample using an ORAGENE kit. Neither participants nor their physicians will receive individual reports of this research. Results will not be placed in the participant's health records. All information will be kept confidential and used only for this research.

There is a rare chance that a research team member could be accidentally exposed to your blood or body fluids. If that occurs, extra blood (about 2 teaspoons) may be drawn to test for infections such as hepatitis and HIV (the AIDS virus). An existing blood sample may be used for these tests instead. You will be told that your blood is being tested and the results of your test. Researchers will ask how you would like to receive the results, such as by phone or certified letter. The test results and your name, address, date of birth, and sex will be recorded in the confidential M. D. Anderson medical records.

If you test positive for hepatitis or HIV, the test results and your name, address, date of birth, and sex will be shared with appropriate health authorities as required by law. You will also be given a list of places in your area so that you can receive further testing and treatment.

For the protection of your privacy, the study staff has obtained a Certificate of Confidentiality from the National Institutes of Health. With this certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the certificate to resist any demands for information that would identify you, except as explained below.

The certificate cannot be used to resist a demand for information from personnel of the United State Government that is used for auditing or evaluation of Federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA).

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the certificate to withhold that information.

This is an investigational study. This study will include a total of 1,000 participants recruited at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1) An effected or uneffected member of a family, age 18 or older, that has two or more reported pancreatic cancers in the family.

Exclusion Criteria:

1. Cases under age 18.
2. Relatives of pancreatic cancer cases under age 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MDACC pancreatic cancer patients and family members (two or more) of someone with pancreatic cancer, all over over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 4770 (Estimated)
Dates: Start 2002-06-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Identification of susceptibility genes in high risk familial pancreatic cancer (FPC) pedigrees using cutting-edge genetic analysis methods | 8 Years
  Data collection from patient response to 30-40 minute questionnaire and blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Daniel-MacDougall, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org